CLINICAL TRIAL: NCT00645437
Title: An Open-Label Randomized Multiple-Dose Study to Evaluate Levofloxacin Steady-State Pharmacokinetics and Safety in Subjects With Varying Degrees of Renal Function
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of Levofloxacin in Patients With Varying Degrees of Renal Function.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004174
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Renal Diseases
Keywords: renal diseases; levofloxacin
MeSH Terms: conditions — Kidney Diseases | interventions — Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin

SUMMARY:
The primary objective was to evaluate the pharmacokinetics and safety of two dosing regimens of levofloxacin in patients with varying degrees of renal function.

DETAILED DESCRIPTION:
In this multiple-dose study conducted at 4 centers, the pharmacokinetics of two dosing regimens of levofloxacin were assessed in medically stable men and women with varying degree of renal function. The study consisted of a 21 day pretreatment screening phase, a 7-day open label treatment phase, and a 7 day posttreatment phase (or a follow-up phase for subjects with early study withdrawal). Patients were randomized into 1 of 10 treatment groups, for a total of 6 patients per group, based on degree of renal function to ensure that creatinine clearance values within each group represented the full range of values defined in the Food and Drug Administration's (FDA) 1998 guideline for pharmacokinetic studies in patients with impaired renal function. Fifty-nine patients were enrolled in the study. All patients received a single 750-mg dose of levofloxacin on Day 1; subsequent doses of either 250, 500, or 750 mg of levofloxacin (q24h or q48h) were based on renal function. Blood samples were collected from each patient from Day 1 to Day 14 for pharmacokinetic evaluation. Urine was collected on Days 1 and 7 before dosing and over specific time intervals up to 24 or 48 hours postdosing depending on the patient's dosing regimen. Dialysate samples were collected on Day 7 from HD patients immediately before dosing (as dialysis began) and at the end of the dialysis treatment. Patients were confined overnight at the study unit on Days 0, 1, 6, and 7, and remained confined until the 24 hour blood samples were collected on Days 2 and 8. Safety was based on the incidence, relationship to therapy, and severity of treatment-emergent adverse events and on changes in clinical laboratory values (hematology, chemistry, and urinalysis), vital sign measurements, electrocardiograms (ECGs), and physical examination findings. Single 750-mg dose of levofloxacin on Day 1; subsequent doses of Levofloxacin 250 milligram (mg), 500 mg, and 750 mg tablets administered every 24 hours for 7 days or every 48 hours for 7 days

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 35 kg/m2
* No prescription or over-the-counter medications for previous 7 days
* Negative tests for drug and alcohol abuse, HIV, hepatitis B and hepatitis C
* Medically stable based on medical history, physical examination, 12-lead electrocardiograms, toxicology, antigen, and antibody screens, and clinical laboratory evaluations
* Stable renal function based on calculated creatine clearance for non-dialysis patients and the same dialysis treatment for at least 6 months prior to screening for dialysis patients
* Patients with creatinine clearance =80 mL/min who require treatment for renal impairment or other chronic disease (e.g., well-controlled diabetes, hypertension) must be on a stable treatment plan (medicines, doses, and regimens) for at least 2 months prior to Day 1 and during the entire study
* Hematocrit (hct) within the normal range based on patients' renal function at screening

Exclusion Criteria:

* Allergic reaction to quinolones
* Known or suspected allergy to heparin
* Clinically significant ECG or clinical laboratory abnormalities
* Creatinine clearance <80 mL/min whose medical condition was unstable
* creatinine clearance >= 80 mL/min who required concomitant medication during the study
* Poorly controlled type 1 or type 2 diabetes
* Patients with creatinine clearance >= 50 mL/min with screening blood pressure outside the normal range (sitting systolic blood pressure <90 or >140 mm mercury [Hg] or diastolic blood pressure <60 or >90 mm Hg)
* Patients with CLCR <50 mL/min who had sitting systolic blood pressure <90 or >160 mm Hg, or diastolic blood pressure <60 or >90 mm Hg
* Required warfarin treatment
* Required immunosuppressive medications for treatment of immune-mediated renal disease or kidney transplant
* Pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pharmacokinetics of two dosing regimens of levofloxacin in renally impaired and dialysis patients.

SECONDARY OUTCOMES:
Safety of two dosing regimens of levofloxacin in renally impaired and dialysis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An Open-Label Randomized Multiple-Dose Study to Evaluate Levofloxacin Steady-State Pharmacokinetics and Safety in Subjects With Varying Degrees of Renal Function — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=560&filename=CR004174_CSR.pdf